CLINICAL TRIAL: NCT03291236
Title: Survival Outcomes of Uterine Cervical Malignancies in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: SOCM-1
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Uterine Cervical Neoplasms; Survival
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Death Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up for death and recurrence of patients — All patients are follow-up to determine specific date of diagnosis, recurrence and death.

SUMMARY:
This study aims to determine survival outcomes (overall survival and progression-free survival) of primary malignancies of uterine cervix in China and relevant risk factors in a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Primary malignancies of uterine cervix.

Exclusion Criteria:

* Secondary malignancies of uternie cervix.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with primary malignancies of uterine cervix in China.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Duration from diagnosis to recurrence
Progression-free survival | 5 years
  Duration from last treatment after remission to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li L, Ma S, Tan X, Zhong S, Wu M. The Urodynamics and Survival Outcomes of Different Methods of Dissecting the Inferior Hypogastric Plexus in Laparoscopic Nerve-Sparing Radical Hysterectomy of Type C: A Randomized Controlled Study. Ann Surg Oncol. 2019 May;26(5):1560-1568. doi: 10.1245/s10434-019-07228-8. Epub 2019 Feb 13. PMID 30759291